CLINICAL TRIAL: NCT02873494
Title: Impedance Cardiography by PhysioFlow® for Non-invasive Cardiac Output Monitoring: a Comparison With Trans-thoracic Echocardiography in Pediatric Intensive Care Patients.
Brief Title: PHYSIOFLOW/Comparison of Cardiac Output Measurement
Acronym: PF-ECHO
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012_25; 2012-A0132835 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-09-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Pediatric Disorders
Keywords: Hemodynamic monitoring; cardiac output; Transthoracic echocardiography; Impedance cardiography; Child; Physioflow; pediatric intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PHYSIOFLOW PF05 Lab1TM: Impedance cardiography
  Interventions: Device: PHYSIOFLOW - PF05 Lab1TM

INTERVENTIONS:
Device: PHYSIOFLOW - PF05 Lab1TM

SUMMARY:
PhysioFlow® (PF®) is a new cardiac output (CO) monitoring method by impedance cardiography (IC), never studied in pediatric intensive care unit (PICU). The aim of the study was to compare CO and cardiac index (CI) measurements (IC) by trans-thoracic Doppler echocardiography (TTE) (COTTE and CITTE) and PF® (COIC and CIIC) in PICU.

DETAILED DESCRIPTION:
In this monocentric prospective study in PICU of the CHRU of Lille, simultaneous sets of three measurements were realized by TTE and PF® in 43 patients.

In the study, the patient will receive a measure of CF by impedancemetry chest. This electrode will be glued on the torso and the neck of the child. We will collect information obtained through IT, to compare the results obtained by the ETT, carried out under the support of the child. The study will last 15 minutes maximum. No blood sampling will be conducted for the purpose of the study, apart from the exams necessary to its support and its treatment. At no time, the results of the impedance will affect support. The study will use only the data contained in the medical file of the child and would involve no additional intervention (no examination, no further treatment). The use of these data will then be anonymous. After anonymization, information recorded will computer processing of the data collected.

Concordance correlation coefficient (CCC) and Bland-Altman analysis with log-transformed data were used to compare CO, CI, stroke volume (SV) and systemic vascular resistance (SVR) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 28 days to 10 years hospitalized in Pediatric ICU, including therapeutic support requires a hemodynamic assessment by ETT.

Exclusion Criteria:

* Refusal of the child or refusal of one of the holders of parental authority
* Cardiac rhythm disorders
* Greater than 240 beats per minute tachycardia
* Burns or skin lesions of thorax
* Poor Echogenicity
* Congenital heart disease complex (except a persistent ductus arterious and interventricular or interventricular communication)
* Aortic insufficiency

Ages: 28 Days to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child hospitalized in pediatric intensive care unit aged from 28 days to 10 years. Any change of treatment was performed during inclusion
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The concordance between DC and IC and SVR measurements obtained with both techniques, IT and the ETT in pediatric intensive care patient. | Within the time hemodynamic assessment by echocardiography, less than 15 minutes.
  The percentage of acceptable error between the two methods must be less than 30%, The aim of the study was to compare CO and cardiac index (CI) measurements by trans-thoracic Doppler echocardiography (TTE) (COTTE and CITTE) and PF® (COIC and CIIC) in PICU.

SECONDARY OUTCOMES:
CO and CI measures | Within the time hemodynamic assessment by echocardiography, less than 15 minutes.
  The concordance of the CO and CI and SVR measures obtained by these two methods in mechanical ventilation and requiring treatments inotropic and vasoactive.

CONTACTS AND LOCATIONS:
Overall Officials: ASTRID BOTTE, PH, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No